CLINICAL TRIAL: NCT00006022
Title: Phase IA/IB Trial of Modulation of the Biological Response to Interleukin-2 (IL-2) With Bryostatin 1 (BRYO; NSC 339555)
Brief Title: Interleukin-2 Plus Bryostatin 1 in Treating Patients With Melanoma or Kidney Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: CDR0000068034; P30CA016059 (NIH); MCV-MCC/CCHR-9910-2A; NCI-T99-0049
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Kidney Cancer; Melanoma (Skin)
Keywords: stage III renal cell cancer; stage IV renal cell cancer; recurrent renal cell cancer; stage III melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Kidney Neoplasms; Melanoma; Carcinoma, Renal Cell | interventions — aldesleukin; bryostatin 1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: aldesleukin
Drug: bryostatin 1

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Interleukin-2 may stimulate a person's white blood cells to kill tumor cells. Combining bryostatin 1 with interleukin-2 may kill more tumor cells.

PURPOSE: Randomized phase I trial to study the effectiveness of interleukin-2 plus bryostatin 1 in treating patients who have melanoma or kidney cancer that cannot be removed during surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the dose of bryostatin 1 that, when administered in conjunction with low-dose interleukin-2, maximizes in vitro interleukin-2- stimulated peripheral blood stem cell proliferation in patients with melanoma or renal cell carcinoma.
* Assess other intermediate markers of immune response in patients treated with this regimen.
* Determine tumor responses, response durations, progression-free intervals, and survival of patients treated with this regimen.

OUTLINE: This is a randomized, double-blind study. Patients are randomized to one of three bryostatin 1 dose levels.

Patients receive interleukin-2 subcutaneously daily on days 1-5 and bryostatin 1 IV over 1 hour on day 1 weekly for 3 weeks. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 21 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed cutaneous or mucosal melanoma or renal cell carcinoma

  * Unresectable disease
* No known uncontrolled CNS metastases

  * CNS metastases allowed only if recently irradiated or known to be controlled

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Hemoglobin at least 8 g/dL
* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3
* Absolute lymphocyte count at least 1,000/mm^3

Hepatic:

* Total bilirubin no greater than 1.5 mg/dL OR
* Conjugated bilirubin no greater than 0.3 mg/dL
* AST no greater than 2.5 times upper limit of normal

Renal:

* Creatinine no greater than 2 mg/dL

Cardiovascular:

* No myocardial infarction within the past 6 months
* No uncontrolled hypertension, angina, or congestive heart failure

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 3 months after study
* No known intolerance to acetaminophen
* No primary or secondary immunodeficiency
* No other condition that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* At least 1 month since prior topical, systemic, or inhaled corticosteroids
* No concurrent topical, systemic, or inhaled corticosteroids

Radiotherapy:

* See Disease Characteristics

Surgery:

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2000-09; Primary Completion 2003-10 (Actual); Study Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D. Roberts, MD, Study Chair — Massey Cancer Center
Locations (2):
- United States (2):
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Massey Cancer Center, Richmond, Virginia